CLINICAL TRIAL: NCT06300970
Title: Efficacy of Artesunate-amodiaquine (ASAQ) and Artemether-lumefantrine (AL) for the Treatment of Uncomplicated Plasmodium Falciparum Malaria in Liberia
Brief Title: Efficacy of Artesunate-amodiaquine and Artemether-lumefantrine for Treatment of Plasmodium Falciparum Malaria in Liberia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Ministry of Health, Liberia (Other)
Responsible Party: Principal Investigator, Jonathan Schultz, Medical Officer, Centers for Disease Control and Prevention
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0900f3eb81e634a9
Record Dates: First submitted 2024-02-13; First posted 2024-03-08 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Plasmodium Falciparum; Malaria; Uncomplicated Malaria
Keywords: Plasmodium falciparum; Anti-malarial therapeutic efficacy study (TES); Artemisinin-based combination therapies (ACT)
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — amodiaquine, artesunate drug combination; Amodiaquine; Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Artesunate+Amodiaquine (ASAQ) (Active Comparator): Amodiaquine-artesunate (ASAQ) dose based on weight, given once daily for three days.
  ASAQ has three formulations, with the dose depending on the weight of the child according to the following.
  4.5-8.9 kg = 1 tablet 25 mg AS/67.5 mg AQ 9-17.9kg = 1 tablet 50 mg AS/135 mg AQ 18.0-35.9kg = 1 tablet 100 mg AS/270 mg AQ
  ≥36.0kg = 2 tablets 100 mg AS/270 mg AQ
  Interventions: Drug: Amodiaquine-artesunate (ASAQ)
- Artemether+Lumefantrine (AL) (Active Comparator): Artemether+Lumefantrine (AL) dose is based on weight and given twice daily for three days. AL has one formulation, with pills containing 20 mg artemether and 120 mg lumefantrine. The number of tablets per dose depends on the weight of the child according to the following:
  5 -14.9 kg = 1 tablet per dose 15 -24.9 kg = 2 tablets per dose 25 -34.9 kg = 3 tablets per dose
  ≥35 kg = 4 tablets per dose
  1 tablet contains 20 mg artemether and 120 mg lumefantrine
  Interventions: Drug: Artemether+Lumefantrine (AL)

INTERVENTIONS:
Drug: Amodiaquine-artesunate (ASAQ) — Oral medication given for treatment of uncomplicated plasmodium falciparum infection.
  Other Names: ASAQ; Camoquin
  Arms: Artesunate+Amodiaquine (ASAQ)
Drug: Artemether+Lumefantrine (AL) — Oral medication given for treatment of uncomplicated plasmodium falciparum infection.
  Other Names: AL; Coartem
  Arms: Artemether+Lumefantrine (AL)

SUMMARY:
To assess the efficacy of both first-line antimalarial medications used for the treatment of uncomplicated Plasmodium falciparum malaria infections in two geographic regions in Liberia.

DETAILED DESCRIPTION:
Title: Efficacy of artesunate+amodiaquine (ASAQ) and artemether+lumefantrine (AL) for the treatment of uncomplicated Plasmodium falciparum malaria in Liberia

Objective: To assess the efficacy of both first-line ASAQ and AL for the treatment of uncomplicated P. falciparum malaria infections

Study Sites: Sacleapea Comprehensive Health Center, Saclepea-Mah District in Nimba County; and Sinje Health Center, Garwula District, Sinje, in Grand Cape Mount County

Study Period: August 2022 to August 2023

Study Design: Prospective study of two cohorts with simultaneous enrolment of each therapy

Patient population: Patients aged 6 to 59 months with confirmed uncomplicated P. falciparum infection

Sample Size: Total number of patients to be enrolled is 352 patients. This consists of 88 patients per arm per site. There are two arms in each of the two sites.

Treatment(s) and follow-up: Patients enrolled in the ASAQ arm will receive the treatment once daily dose for three days. Patients enrolled in the AL arm will receive treatment twice daily dose for three days. Clinical and parasitological parameters will be monitored over a 28-day follow-up period to evaluate drug efficacy.

Primary endpoints: The proportion of patients with early treatment failure, late clinical failure, late parasitological failure or an adequate clinical and parasitological response as indicators of efficacy. Recrudescence will be distinguished from re-infection by polymerase chain reaction (PCR) analysis.

Secondary endpoints: The frequency and nature of adverse events will be recorded.

Exploratory endpoints: Any polymorphisms of molecular markers for antimalarial drug resistance and prevalence of HRP2 deletions.

ELIGIBILITY:
Inclusion Criteria

1. Age between 6 to 59 months (5 years)
2. Weight ≥ 5 kg
3. Monoinfection with P. falciparum with a parasite density of 2,000 to 200,000 asexual forms per microliter of blood
4. Axillary temperature ≥37.5˚C or history of fever in the last 24 hours
5. Hemoglobin ≥ 8.0g/dl
6. Easy access to the health facility and ability to return to the health facility over the course of the four weeks of follow-up
7. Informed consent of parent or guardian

Exclusion Criteria on Day 0

1. Any danger signs or signs of severe malaria (see Appendix I)
2. Pneumonia or bronchopneumonia
3. Severe malnutrition (Z-score < 3)
4. History of taking antimalarials (or antibiotics with antimalarial activity such as cotrimoxazole, tetracycline or doxycycline) in the last 14 days
5. Mixed malaria infection
6. History of hypersensitivity or allergy to the medication

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 352 (Actual)
Dates: Start 2022-08-09 (Actual); Primary Completion 2023-08-16 (Actual); Study Completion 2023-08-16 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Early Treatment Failure (ETF) | Day 1 to day 3 following treatment.
  * Danger signs or severe malaria on day 1, 2, or 3 in the presence of parasitemia
  * A parasitemia on day 2 higher than day 0
  * Axillary temperature ≥ 37.5 °C on day 3 in the presence of parasitemia
  * Parasitemia on day 3 ≥ 25% of day 0 parasitemia
Number of Participants with Late Treatment Failure (LTF) | Day 4 to day 28 following treatment.
  * Danger signs, signs of severe malaria, or axillary temperature > 37.5 °C in the presence of parasitemia on any day between day 4 and day 28 in patients who did not previously meet any of the criteria of early treatment failure
  * Presence of parasitemia (with a parasite with the same genotype as day 0) on any day between day 7 and day 28 regardless of temperature in patients who did not previously meet any of the criteria of early treatment failure
Number of Participants with Adequate Clinical and Parasitological Response (APCR) | Day 28 following treatment.
  • Absence of parasitemia on day 28, irrespective of axillary temperature, in patients who did not previously meet any of the criteria of early treatment failure, late clinical failure, reinfection or late parasitological failure.

SECONDARY OUTCOMES:
Number of Patients with Adverse Events | During participation in the study, approximately 4 weeks.
  An adverse event is defined as any unfavorable, unintended sign, symptom, syndrome or disease that develops or worsens with the use of a medicinal product, regardless of whether it is related to the medicinal product during participation in the study, approximately 4 weeks.

OTHER OUTCOMES:
Number of samples with confirmed Histidine-rich protein 2/3 (HRP2/3) gene deletions | Samples collected from participants during the study, approximately 4 weeks.
  Molecular data on hrp2/hrp3 deletions will be tabulated and frequencies will be calculated from samples collected during the study, approximately 4 weeks.
Number of samples with molecular markers of anti-malarial resistance | Samples collected from participants during the study, approximately 4 weeks.
  Molecular data on drug resistance polymorphisms will be tabulated and frequencies will be calculated from samples collected during the study, approximately 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Victor S Koko, Principal Investigator — Liberia National Malaria Control Program
Locations (2):
- Liberia (2):
  - Sinje Health Center, Garwula District, Sinje, Grand Cape Mount County, Sinje, Grand Cape Mount County
  - Saclepea-Mahn Comprehensive Health Center Saclepea-Mahn District, Nimba County, Saclepea, Nimba

IPD SHARING:
Plan to Share IPD: Yes
IPD should be requested from the Liberian Ministry of Health
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Supporting information and data can be requested from the Liberian Ministry of Health.
Access Criteria: Supporting information and data can be requested from the Liberian Ministry of Health.